CLINICAL TRIAL: NCT07402291
Title: Comparative Effects of Mulligan's Pain Release Phenomenon and Kaltenborn Mobilizations on Pain, Range of Motion And Disability in Patients With Knee Osteoarthritis.
Brief Title: Effects of Mulligan's Pain Release Phenomenon and Kaltenborn Mobilizations on Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0199
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthritis
Keywords: Manual Therapy; Manual Mobilization; Disabilty; Convectional Exercises; Range of Motion
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Traction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan's pain release phenomenon (Experimental): 22 participants were allocated into Experimental group A, Mulligans Pain release compression were performed for 5 repetitions with 20-30 seconds hold with 5 seconds rest. Convectional treatment included hot pack for 10 mins and ultrasound for 8 mins. Exercises includes stretches for Hamstring, Gastrocnemius, Soleus and Rectus femoris for 3 set with 10 repetitions and 10 seconds hold. Quadricep setting exercise, Full arc extension and Straight leg raises was done for 1 set of 10 repetitions and cycling was performed for 2 minutes. A total of 18 sessions were conducted for 6 weeks with 3 sessions scheduled every week. Outcome measures were measured in week 1 before the treatment and after 6 weeks of treatment.
  Interventions: Other: Mulligan's pain release phenomenon
- Kaltenborn mobilization with traction (Experimental): 22 participants were allocated into Experimental group B, Kaltenborn grade III mobilization with traction were performed for 10 repetitions with 3 sets treatment included hot pack for 10 mins and ultrasound for 8 mins. Exercises includes stretches for Hamstring, Gastrocnemius, Soleus and Rectus femoris for 3 set with 10 repetitions and 10 seconds hold. Quadricep setting exercise, Full arc extension and Straight leg raises was done for 1 set of 10 repetitions and cycling was performed for 2 minutes. A total of 18 sessions were conducted for 6 weeks with 3 sessions scheduled every week. Outcome measures were measured in week 1 before the treatment and after 6 weeks of treatment.
  Interventions: Other: Kaltenborn mobilization with traction

INTERVENTIONS:
Other: Mulligan's pain release phenomenon — Experimental Group A was given Mulligan's pain release phenomenon compression techniques along with conventional therapy for 3 sessions per week for 6 weeks in total. After Hot pack for 10 mins and Ultrasound for 8 mins participants performed series of exercises included targeted muscles stretchings (Hamstrings, Quadriceps, Soleus and Rectus femoris) 10 repetitions x 3 sets and 10 seconds hold. Quadricep setting exercise, Full arc extension and Straight leg raises for 10 repetitions x 1 set followed by cycling for 2 mins.
  Arms: Mulligan's pain release phenomenon
Other: Kaltenborn mobilization with traction — Experimental Group b was given grade III Kaltenborn mobilization with traction along with conventional therapy for 3 sessions per week for 6 weeks in total. After Hot pack for 10 mins and Ultrasound for 8 mins participants performed series of exercises included targeted muscles stretchings (Hamstrings, Quadriceps, Soleus and Rectus femoris) 10 repetitions x 3 sets and 10 seconds hold. Quadricep setting exercise, Full arc extension and Straight leg raises for 10 repetitions x 1 set followed by cycling for 2 mins.
  Arms: Kaltenborn mobilization with traction

SUMMARY:
Knee osteoarthritis is a degenerative condition that is prevalent in older population and is associated with pain, stiffness, decreased range of motion and impaired function. Physical therapy techniques, such as Mulligan's Pain Release Phenomenon and Kaltenborn Mobilization are used to alleviate patient's symptoms.

A Randomized Clinical Trial was conducted at SAP Rehab Center (Saira Memorial hospital) and Pak Health Care, Lahore. 44 participants age between 40-65 years with Knee Osteoarthritis were randomly assigned into 2 groups. Both groups underwent treatment three times a week for total of six weeks. Group A received treatment through Mulligan's Pain Release Phenomenon along with conventional exercises. Group B received treatment through Kaltenborn mobilization and conventional exercises. Convectional treatment started with hot pack for 10 minutes followed by ultrasound for 8 minute, the program indcluded a series of exercises (Hamstring stretch, Gastrocnemius Stretch, Soleus Stretch and Rectus femoris Stretch all for 3 set with 10 repetitions and 10 seconds hold. Quadricep setting exercises 1 set with 10 repetitions, Full arc extension and Straight leg raises 1 set and 10 repetitions. the exercises program ended with cycling for 2 minutes. Outcome measures were conducted through NPRS for pain, WOMAC for functional disability, Universal Goniometer for range of motion at baseline and after 6 weeks. Data was analyzed through SPSS software version 27.

The aim of the study is to compare the effects of Mulligan's Pain Release Phenomenon and Kaltenborn Mobilization on pain, disability and range of motion in patients with early Knee Osteoarthritis.

DETAILED DESCRIPTION:
The objective of my study is to determine the comparative effects of Mulligan's Pain Release Phenomenon and Kaltenborn Mobilization on pain, disability and range of motion in patients with early Knee Osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age included between 40-65 years
* NPRS pain rating above 3
* Both Genders
* Diagnosed with Grade 1 and Grade 2 knee osteoarthritis
* Unilateral knee pain
* Pain for more than 3 months
* Decrease range of motion

Exclusion Criteria:

* Age more than 60 years
* Bilateral knee pain
* Patellofemoral pain syndrome
* Rheumatoid Arthritis
* Fracture or ligamentous injury of lower extremity
* Any trauma, burn, infection or tumor around the knee
* Total knee replacement

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6 weeks
  The Numeric Pain Rating Scale is a uni dimensional measure of pain severity in adults, including those with chronic pain caused by rheumatic disorders. It is a 11 point numeric scale ranging from "0" representing no pain and "10" worst pain possible. In this questionnaire the respondent selects a whole number from 0-10 that best reflects their intensity of pain, 1-3 means mild pain, 4-6 indicates moderate and 7-10 means severe pain.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 weeks
  Western Ontario and McMaster Universities Osteoarthritis Index is widely used is evaluation of hip and knee osteoarthritis. This questionnaire have 24 items with 3 sub scales, measure pain (5 items), stiffness (2 items) and and physical function (17 items).
ROM Knee (Flexion) | 6 weeks
  Change from Baseline ROM of Knee Flexion was taken with the help of Universal Goniometer
ROM Knee (Extension) | 6 weeks
  Change from Baseline ROM of Knee Extension was taken with the help of Universal Goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Ameena Amjad, Ph.D, Principal Investigator — Riphah International University
Locations (1):
- SAP Rehab Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taj S, Anwar K, Arshad H, Khalid M, Ali MQ, Hussain E. Effectiveness of Maitland Mobilization versus Pain release phenomena for pain, range of motion and disability in early knee osteoarthritis. Pakistan Journal of Medical & Health Sciences. 2023;17(01):30-.
- [Background] Bacon K, LaValley MP, Jafarzadeh SR, Felson D. Does cartilage loss cause pain in osteoarthritis and if so, how much? Ann Rheum Dis. 2020 Aug;79(8):1105-1110. doi: 10.1136/annrheumdis-2020-217363. Epub 2020 May 7. PMID 32381567
- [Background] Sherazi F, Waqar S, Khalid M, Saleem K, Kiani SK, Shahzad M. Effect of knee joint mobilization on hamstring muscle length in patient with knee osteoarthritis. The Rehabilitation Journal. 2022;6(04):468-73.
- [Background] Abramoff B, Caldera FE. Osteoarthritis: Pathology, Diagnosis, and Treatment Options. Med Clin North Am. 2020 Mar;104(2):293-311. doi: 10.1016/j.mcna.2019.10.007. Epub 2019 Dec 18. PMID 32035570
- [Background] Olsson S, Akbarian E, Lind A, Razavian AS, Gordon M. Automating classification of osteoarthritis according to Kellgren-Lawrence in the knee using deep learning in an unfiltered adult population. BMC Musculoskelet Disord. 2021 Oct 2;22(1):844. doi: 10.1186/s12891-021-04722-7. PMID 34600505
- [Background] Callahan LF, Cleveland RJ, Allen KD, Golightly Y. Racial/Ethnic, Socioeconomic, and Geographic Disparities in the Epidemiology of Knee and Hip Osteoarthritis. Rheum Dis Clin North Am. 2021 Feb;47(1):1-20. doi: 10.1016/j.rdc.2020.09.001. Epub 2020 Oct 29. PMID 34042049
- [Background] Berteau JP. Knee Pain from Osteoarthritis: Pathogenesis, Risk Factors, and Recent Evidence on Physical Therapy Interventions. J Clin Med. 2022 Jun 7;11(12):3252. doi: 10.3390/jcm11123252. PMID 35743322
- [Background] Xie R, Yao H, Mao AS, Zhu Y, Qi D, Jia Y, Gao M, Chen Y, Wang L, Wang DA, Wang K, Liu S, Ren L, Mao C. Biomimetic cartilage-lubricating polymers regenerate cartilage in rats with early osteoarthritis. Nat Biomed Eng. 2021 Oct;5(10):1189-1201. doi: 10.1038/s41551-021-00785-y. Epub 2021 Oct 4. PMID 34608279
- [Background] Sanchez-Lopez E, Coras R, Torres A, Lane NE, Guma M. Synovial inflammation in osteoarthritis progression. Nat Rev Rheumatol. 2022 May;18(5):258-275. doi: 10.1038/s41584-022-00749-9. Epub 2022 Feb 14. PMID 35165404
- [Background] Hendrika W, Reswari A. The effect of physiotherapy on pain improvement in patients with early knee osteoarthritis at RSU UKI. International Journal of Medical and Health Research. 2021;7(6):52-9.
- [Background] Ozden F, Nadiye Karaman O, Tugay N, Yalin Kilinc C, Mihriban Kilinc R, Umut Tugay B. The relationship of radiographic findings with pain, function, and quality of life in patients with knee osteoarthritis. J Clin Orthop Trauma. 2020 Jul;11(Suppl 4):S512-S517. doi: 10.1016/j.jcot.2020.04.006. Epub 2020 Apr 9. PMID 32774020
- [Background] Geng R, Li J, Yu C, Zhang C, Chen F, Chen J, Ni H, Wang J, Kang K, Wei Z, Xu Y, Jin T. Knee osteoarthritis: Current status and research progress in treatment (Review). Exp Ther Med. 2023 Aug 25;26(4):481. doi: 10.3892/etm.2023.12180. eCollection 2023 Oct. PMID 37745043
- [Background] Elboim-Gabyzon M, Nahhas F. Laser therapy versus pulsed electromagnetic field therapy as treatment modalities for early knee osteoarthritis: a randomized controlled trial. BMC Geriatr. 2023 Mar 16;23(1):144. doi: 10.1186/s12877-022-03568-5. PMID 36922781
- [Background] Umar M, Anwar A, Khan N, Marryam M, Rashid H. Effectiveness Of Kaltenborn Mobilization Versus Muscle Energy Technique On Shoulder Range Of Motion In Adhesive Capsulitis. Journal of Rawalpindi Medical College. 2023;27(3).
- [Background] Anwar S, Javaid M, Malik S, Asghar MU, Perveen W, Chaudary M. Effects of mulligan pain release phenomenon technique in management of patellofemoral pain syndrome: RCT. Pakistan Journal of Medical & Health Sciences. 2022;16(03):72-.
- [Background] Bhagat M, Neelapala YVR, Gangavelli R. Immediate effects of Mulligan's techniques on pain and functional mobility in individuals with knee osteoarthritis: A randomized control trial. Physiother Res Int. 2020 Jan;25(1):e1812. doi: 10.1002/pri.1812. Epub 2019 Sep 10. PMID 31502354
- [Background] Lalnunpuii A, Sarkar B, Alam S, Equebal A, Biswas A. Efficacy of mulligan mobilisation as compared to Maitland mobilisation in females with knee osteoarthritis: a double blind randomized controlled trial. International Journal of Therapies and Rehabilitation Research. 2017;6(2):37.
- [Background] Mangus BC, Hoffman LA, Hoffman MA, Altenburger P. Basic principles of extremity joint mobilization using a Kaltenborn approach. Journal of Sport Rehabilitation. 2002;11(4):235-50.